CLINICAL TRIAL: NCT04549025
Title: Phase 2 Study of PD-1 Inhibitor JTX-4014 Alone and in Combination With Vopratelimab, an ICOS Agonist, in Biomarker-selected Subjects With Metastatic NSCLC After One Prior Platinum-containing Regimen
Brief Title: Study of PD-1 Inhibitor JTX-4014 Alone and in Combination With Vopratelimab in Biomarker-selected Subjects With Metastatic NSCLC After One Prior Platinum-containing Regimen
Acronym: SELECT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor decided to discontinue development of pimivalimab prior to the planned study completion. At the time of the decision to discontinue development, enrollment in the study had been completed.
Sponsor: Jounce Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JTX-4014-202
Record Dates: First submitted 2020-09-01; First posted 2020-09-16 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Monotherapy Cohort 1 (MC1) (Experimental): Enrolled patients will receive 1000 mg pimivalimab (JTX-4014) administered alone every 6 weeks (q6w).
  Interventions: Drug: Pimivalimab
- Combination Therapy Cohort 1 (CC1) (Experimental): For Cycle 1, enrolled patients will receive 0.1 mg/kg vopratelimab (JTX-2011) on Day 1, followed by 1000 mg pimivalimab (JTX-4014) on Day 8. For Cycle 2 and beyond, vopratelimab and pimivalimab will be administered in combination (on Day 1) q6w.
  Interventions: Drug: Pimivalimab; Drug: Vopratelimab
- Combination Therapy Cohort 2 (CC2) (Experimental): For Cycle 1, enrolled patients will receive 0.03 mg/kg vopratelimab (JTX-2011) on Day 1, followed by 1000 mg pimivalimab (JTX-4014) on Day 8. For Cycle 2 and beyond, vopratelimab and pimivalimab will be administered in combination (on Day 1) q6w.
  Interventions: Drug: Pimivalimab; Drug: Vopratelimab

INTERVENTIONS:
Drug: Pimivalimab — Specified dose on specified days
  Other Names: JTX-4014
Drug: Vopratelimab — Specified dose on specified days
  Other Names: JTX-2011
  Arms: Combination Therapy Cohort 1 (CC1); Combination Therapy Cohort 2 (CC2)

SUMMARY:
This is a Phase 2, open-label study to evaluate PD-1 inhibitor pimivalimab (JTX-4014) alone and in combination with vopratelimab (JTX-2011), an ICOS agonist, in biomarker-selected adult subjects with metastatic NSCLC who are PD-1/PD-L1 inhibitor naïve and have progressed on a platinum-based chemotherapy regimen.

DETAILED DESCRIPTION:
Pimivalimab is a fully human IgG4 monoclonal antibody designed to specifically bind to programmed cell death receptor protein-1 (PD-1) and block its interaction with its ligands, programmed cell death receptor protein-1 ligand 1 (PD-L1) and programmed cell death receptor protein-1 ligand 2 (PD-L2), to augment anti-tumor T cell activity. Vopratelimab is an agonist monoclonal antibody that specifically binds to the Inducible CO-Stimulator of T cells (ICOS) to generate an anti-tumor immune response. This is a Phase 2, open label study to evaluate the efficacy, safety, tolerability of pimivalimab alone and in combination with vopratelimab in biomarker-selected adult subjects with metastatic non-small cell lung cancer (NSCLC) who are PD-1/PD-L1 inhibitor naïve and have progressed on a platinum-based chemotherapy regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to participate and comply with all study requirements and provide signed and dated informed consent prior to initiation of any study procedures;
2. Histologically or cytologically confirmed diagnosis of NSCLC with evaluable or measurable disease according to RECIST v1.1 with at least 1 measurable lesion;
3. Confirmed tumor RNA signature score in accordance with the study protocol;
4. Previously treated for locally advanced or metastatic NSCLC with 1 prior systemic antineoplastic platinum-containing regimen. Regimen should consist of chemotherapy or with bevacizumab;
5. Age of ≥18 years;
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
7. Predicted life expectancy of ≥ 3months;
8. Specified laboratory values in accordance with the study protocol;
9. If with medical history of the following, eligibility should be discussed with the Medical Monitor:

   1. Prior biliary tract disorders (based on Medical Dictionary for Regulatory Activities [MedDRA] system organ class of Hepatobiliary disorders and MedDRA high-level terms of Obstructive bile duct disorders, Hepatic vascular disorders, and Structural and other bile duct disorders);
   2. Portal hypertension and/or hepatic vascular disorders;
10. For women of childbearing potential (WOCBP): negative serum pregnancy test within 72 hours prior to planned Cycle 1, Day 1 (C1D1) and a negative urine or serum pregnancy test on C1D1. In addition, the WOCBP must be willing to complete a urine or serum pregnancy test prior to each dose of either study drug;
11. WOCBP and males whose partners are WOCBP must agree to use a highly effective method of birth control throughout their participation and for 5 months following the last study drug administration. Highly effective methods of birth control are defined as those that, alone or in combination, result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly.

Exclusion Criteria:

1. Concurrent anticancer treatment or subject is expected to require any other form of antineoplastic therapy while on study, either approved or investigational;
2. Current or past participation in a study of an investigational agent or using an investigational device in the metastatic setting;
3. Chemotherapy <28 days prior to planned C1D1
4. Prior immunotherapy including, but not limited to PD-1 or PD-L1 inhibitor monoclonal antibody (mAb) at any time, including pimivalimab; therapy with any mAb that specifically binds to ICOS, including vopratelimab; or chimeric antigen receptor T cell therapy;
5. Organ transplantation, including allogenic or autologous stem cell transplantation;
6. Use of anticancer therapies listed below in the metastatic setting (allowed as prior treatment for localized disease):

   1. Biologic therapy
   2. Targeted therapy, with the exception of bevacizumab if administered in combination with a platinum-based chemotherapy regimen as first line treatment
7. Positive test for any of the following epidermal growth factor receptor gene mutations in blood or tumor: Exon 18 G719A; Exon 18 G719C; Exon 18 G719S; Exon 19 Del; Exon 20 S768I; Exon 20 T790M; Exon 20 Ins; Exon 21 L858R; Exon 21 L861Q;
8. The following toxicity history:

   1. Ongoing toxicity attributed to prior therapy that was Grade >1 according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE); Exceptions: Grade >1 toxicities that, in the opinion of the Investigator, should not exclude the subject (e.g., alopecia, Grade 2 neuropathy, hypo- or hyperthyroidism, or other endocrinopathies that are well controlled with hormone replacement therapy) and are approved by the Medical Monitor;
   2. History of pneumonitis or interstitial lung disease;
   3. Symptomatic ascites or pleural effusion (subjects who are clinically stable for >3 months following treatment for these conditions [including therapeutic thoraco- or paracentesis] are eligible);
   4. If with medical history of the following, eligibility should be discussed with the Medical Monitor: colitis, hepatitis, nephritis, skin reactions, or encephalitis;
9. Known severe intolerance or life-threatening hypersensitivity reactions to humanized mAbs or IV Ig preparations; any history of anaphylaxis; prior history of human anti-human antibody response; or known allergy to any of the study drugs (including their analogues or excipients [L-Histidine, mannitol, sodium chloride, or polysorbate 80]);
10. Major surgery (excluding minor procedures, e.g., placement of vascular access, gastrointestinal/biliary stent, and biopsy) < 4 weeks prior to planned C1D1;
11. Prior whole brain radiation;
12. Subjects with the following should be reviewed with the Medical Monitor prior to enrollment:

    1. Brain metastases, leptomeningeal disease, or spinal cord compression not definitively treated with surgery or radiation;
    2. Radiation (other than whole brain radiation) has been or will be administered <21 days prior to planned C1D1;
13. Active and clinically relevant bacterial, fungal, or viral infection, including known hepatitis B, C, or human immunodeficiency virus (testing not required);
14. Women who are pregnant, breastfeeding, or who plan to become pregnant/breastfeed while on study; men who plan to father children during the study;
15. Concurrent second malignancy;
16. An active autoimmune disease or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents at a dose of ≥10 mg/day of prednisone equivalent. Subjects who require intermittent use of bronchodilators or local steroid injections will not be excluded from the study. Subjects with hypothyroidism who are stable on hormone replacement therapy will not be excluded from the study;
17. Medical or social condition that, in the opinion of the Investigator, might place the subject at an increased risk, adversely affect compliance, or confound safety or other clinical study data interpretation;
18. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2024-04-25 (Actual)

PRIMARY OUTCOMES:
Change in measurable lesion size | over 9 and 18 weeks (average)
  Mean percent change from baseline tumor size of all measurable existing and new lesions

SECONDARY OUTCOMES:
Overall response rate (ORR) | up to 24 months
  ORR (percentage of subjects with complete response [CR] + partial response [PR]) according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Progression-free survival (PFS) | up to 24 months
  PFS according to RECIST v1.1
Landmark PFS rate | 9 months
  Landmark PFS rate at 9 months according to RECIST v1.1
Disease control rate (DCR) | up to 24 months
  DCR (confirmed CR + confirmed PR + unconfirmed stable disease [SD]) according to RECIST v1.1
Duration of response (DOR) | up to 24 months
  DOR in months according to RECIST v1.1
Overall survival (OS) | up to 24 months
Treatment-emergent adverse events (TEAEs) | up to 24 months
  Incidence and grade of TEAEs
Pharmacokinetic properties of pimivalimab and vopratelimab - Cmax (maximum observed concentration) | Cycle 1 through Cycle 6 (each cycle is 6 weeks)
Pharmacokinetic properties of pimivalimab and vopratelimab - Tmax (time of first occurrence of Cmax) | Cycle 1 through Cycle 6 (each cycle is 6 weeks)
Pharmacokinetic properties of pimivalimab and vopratelimab - AUClast (area under the concentration-time curve from time zero to the last measurable concentration) | Cycle 1 through Cycle 6 (each cycle is 6 weeks)
Pharmacokinetic properties of pimivalimab and vopratelimab - half-life (time it takes for the concentration of the drug in the plasma or the total amount in the body to be reduced by 50%) | Cycle 1 through Cycle 6 (each cycle is 6 weeks)
Pharmacokinetic properties of pimivalimab and vopratelimab - clearance (efficiency of drug elimination) | Cycle 1 through Cycle 6 (each cycle is 6 weeks)
Pharmacokinetic properties of pimivalimab and vopratelimab - volume of distribution (amount of drug in the body divided by the plasma drug concentration) | Cycle 1 through Cycle 6 (each cycle is 6 weeks)
Incidence of anti-drug antibodies (ADAs) to either pimivalimab or vopratelimab | Cycle 1 through Cycle 6 (each cycle is 6 weeks)
Incidence of neutralizing antibodies (NAbs) to either pimivalimab or vopratelimab | Cycle 1 through Cycle 6 (each cycle is 6 weeks)
Association of baseline tumor RNA signature score with clinical outcomes | up to 24 months
  Change in measurable lesion size for patients with elevated tumor RNA signature score (i.e., tumor inflammation signature (TIS) vopra score ≥ 7.9)

CONTACTS AND LOCATIONS:
Overall Officials: Stew Kroll, Study Director — Jounce Therapeutics, Inc.
Locations (72):
- Belarus (2):
  - Minsk City Clinical Oncology Dispensary, Minsk
  - N. N. Alexandrov National Cancer Centre, Minsk
- Bosnia and Herzegovina (2):
  - University Clinical Center of the Republic of Srpska, Banja Luka
  - Clinical Center University of Sarajevo, Sarajevo
- Bulgaria (5):
  - Multiprofile Hospital for Active Treatment - Dobrich AD, Dobrich
  - Multiprofile Hospital for Active Treatment - Uni Hospital OOD, Panagyurishte
  - Complex Oncology Center Plovdiv, Plovdiv
  - Acibadem City Clinic Multiprofile Hospital for Active Treatment Tokuda, Sofia
  - Multiprofile Hospital for Active Treatment Serdika EOOD, Sofia
- Croatia (4):
  - Clinical Hospital Centre Osijek, Osijek
  - General Hospital Pula, Pula
  - University Hospital of Split, Split
  - Klinicki bolnicki centar Zagreb, Zagreb
- Arensia Tbilisi - PPDS, Tbilisi, Georgia
- Hungary (3):
  - Veszprem Megyei Tudogyogyintezet, Farkasgyepű
  - Bács-Kiskun Varmegyei Oktatokorhaz, Kecskemét
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Latvia (2):
  - Pauls Stradins Clinical University Hospital, Riga
  - Riga East Clinical University Hospital, Latvian Oncology Center, Riga
- Arensia Chisinau - PPDS, Chisinau, Moldova
- Romania (4):
  - Affidea Romania SRL, Bucharest
  - Prof Dr I Chiricuta Institute of Oncology, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Sf. Apostol Andrei Constanta, Constanța
  - Oncology Center Sfantul Nectarie, Craiova
- Russia (17):
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk
  - Chelyabinsk Regional Clinical Oncology Dispensary, Chelyabinsk
  - Republican Clinical Oncology Dispensary of Ministry of Healthcare of Tatarstan Republic, Kazan'
  - Krasnoyarsk Regional Oncology Center n.a. A.I. Kryzhanovskiy, Krasnoyarsk
  - Kursk Regional Oncology Centre, Kursk
  - Vitamed Multidisciplinary Medical Center, Moscow
  - Nizhniy Novgorod City Oncology Center, Nizhny Novgorod
  - Clinical Oncology Dispensary, Omsk
  - PMI Euromedservice, Pushkin
  - Ryazan State Medical University n.a. I.P. Pavlov, Ryazan
  - First St. Petersburg State Medical University n.a. I.P Pavlov, Saint Petersburg
  - GBUZ St. Petersburg Clinical Research Center of Specialized Types of Care Oncology n.a. Napalkova, Saint Petersburg
  - JSC "Current medical technologies", Saint Petersburg
  - Mordovia State University, Saransk
  - Research Oncology Institute of Tomsk Scientific Center, Tomsk
  - Volgograd Regional Clinical Oncology Dispensary, Volgograd
  - Regional Clinical Oncology Hospital, Yaroslavl
- Serbia (5):
  - Clinical Hospital Center Bezanijska Kosa, Belgrade
  - Institute for Oncology and Radiology of Serbia - PPDS, Belgrade
  - University Clinical Center of Serbia - PPDS, Belgrade
  - Institute of Lung Diseases Vojvodina, Kamenitz
  - University Clinical Center Kragujevac, Kragujevac
- Slovakia (2):
  - Narodny onkologicky - PPDS, Bratislava
  - Vychodoslovensky onkologicky ustav, a.s., Košice
- Turkey (Türkiye) (9):
  - Adana Sehir Egitim ve Arastirma Hastanesi, Adana
  - Hacettepe University Medical Faculty Hospital, Ankara
  - Akdeniz University Medical Faculty Hospital, Antalya
  - Trakya Universitesi Saglik Arastirma ve Uygulama Merkezi Hastane - Hematoloji Bilim Dali, Edirne
  - Istanbul University Cerrahpasa Medical Faculty Hospital, Istanbul
  - T.C. Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
  - Izmir Ekonomi University Medical Point Hospital, Izmir
  - Inonu University Faculty of Medicine Turgut Ozal Medical Center, Malatya
- Ukraine (15):
  - Communal Nonprofit Enterprise Clinical Center of Oncology, Hematology, Transplantology and Palliative Care of ChOC, Cherkasy
  - Communal Nonprofit Enterprise City Clinical Hospital #4 of Dnipro City Council, Dnipro
  - Municipal Nonprofit Enterprise SubCarpathian Clinical Oncological Centre of Ivano-Frankivsk RC, Ivano-Frankivsk
  - Arensia Kapitanivka - PPDS, Kapitanivka
  - Communal Nonprofit Enterprise Regional Center of Oncology, Kharkiv
  - SI Institute of Medical Radiology and Oncology n.a. S.P. Hryhoriev of NAMS of Ukraine, Kharkiv
  - Communal Nonprofit Enterprise Khmelnytskyi Regional Antitumor Center of Khmelnytskyi Regional Council, Khmelnytskyi
  - Private Enterprise Private Manufacturing Company Acinus, Kropyvnytskyi
  - Clinic of National Institute of Cancer, Kyiv
  - Communal Nonprofit Enterprise Kyiv City Clinical Oncological Center, Kyiv
  - Kyiv Railway Clinical Hospital #3 of Branch Health Center of the PJSC Ukrainian Railway, Kyiv
  - Medical Center of LLC ARENSIA Exploratory Medicine, Kyiv
  - ME Volyn Regional Clinical Hospital of the Volyn Regional Council Regional Medical Oncology Centre, Lutsk
  - Medical and diagnostic center of MediX-Ray International Group LLC Israeli Oncology Hospital LISOD, Obukhiv
  - MNPE Central City Clinical Hospital of Uzhhorod City Council, Uzhhorod